CLINICAL TRIAL: NCT01873508
Title: A Single-center, Open Label, Randomized Cross-over Study to Compare 3 Modified-release Formulations With Different Release Profiles of RO4917523 Along With a Reference Intravenous Microdose Infusion
Brief Title: A Study of Three Modified-Release Formulations of RO4917523 in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None
Other Study IDs: NP28738; 2013-000502-28 (EudraCT Number)
Record Dates: First submitted 2013-06-06; First posted 2013-06-10 (Estimated); Last update posted 2015-09-10 (Estimated); Status verified 2015-09

CONDITIONS: Healthy Volunteer
MeSH Terms: interventions — 2-chloro-4-(1-(4-fluorophenyl)-2,5-dimethyl-1H-imidazol-4-ylethynyl)pyridine

ARMS (3):
- Fast release MR capsule (Experimental)
  Interventions: Drug: RO4917523
- Slow release MR capsule (Experimental)
  Interventions: Drug: RO4917523
- Target release MR capsule (Experimental)
  Interventions: Drug: RO4917523

INTERVENTIONS:
Drug: RO4917523 — Fast release MR capsule, single dose
  Arms: Fast release MR capsule
Drug: RO4917523 — Target release MR capsule, single dose
  Arms: Target release MR capsule
Drug: RO4917523 — Slow release MR capsule, single dose
  Arms: Slow release MR capsule
Drug: RO4917523 — [13C]-labeled tracer dose i.v.
  Arms: Target release MR capsule

SUMMARY:
This single-center, open label, randomized, 3-period cross-over study will compare 3 modified-release formulations of RO4917523 in healthy volunteers. Subjects will be randomized to one of six sequences to receive single oral doses of RO4917523 slow, target and fast release modified release (MR) capsules along with a reference intravenous microdose with the target capsule. A washout period of at least 21 days will occur between treatments.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male and female volunteers, 18 - 55 years of age inclusive Healthy status will be defined by absence in evidence of any active or chronic disease following a detailed medical and surgical history and a complete physical examination
* Body mass index (BMI) of 18 to 30 kg/m2, inclusive, and body weight of at least 50 kg
* Females of child-bearing potential must agree to use effective contraception as defined by protocol
* Non-smoker for at least 90 days prior to dosing on Day 1

Exclusion Criteria:

* History or presence of a clinically significant psychiatric condition as defined by protocol
* Participation in an clinical study with an investigational drug within 60 days or 5 times the half-life (whichever is longer) preceding first administration of study drug. Participation in more than 3 other drug studies within 10 months preceding first administration of study drug.
* Clinically significant disease or disorder
* Personal or family history of long QT syndrome or sudden death
* Any suspicion or history of alcohol and/or other substance abuse or dependence in the last 6 months
* Subject likely to need concomitant medication during the study (including for dental conditions), except for hormonal contraception or HRT
* Pregnant or lactating women, or women who intend to become pregnant during the course of the study
* Positive for hepatitis B, hepatitis C or HIV infection
* Any confirmed significant allergic reactions against any drug, or multiple allergies

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2013-06; Primary Completion 2013-08 (Actual); Study Completion 2013-08 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetics: Area under the concentration-time curve (AUC) | Pre-dose and up to 144 hours post-dose
Pharmacokinetics: Maximum concentration (Cmax) | Pre-dose and up to 144 hours post-dose

SECONDARY OUTCOMES:
Pharmacokinetics: Time to maximum plasma concentration (tmax) | Pre-dose and up to 144 hours post-dose
Pharmacokinetics: Elimination half-life (t1/2) | Pre-dose and up to 144 hours post-dose
Pharmacokinetics: Elimination rate constant: (kel) | Pre-dose and up to 144 hours post-dose
Pharmacokinetics: Absolute bioavailability (F) | Pre-dose and up to 144 hours post-dose
Pharmacokinetics: Total body clearance (CL) | Pre-dose and up to 144 hours post-dose
Pharmacokinetics: Volume of distribution (Vd) | Pre-dose and up to 144 hours post-dose
Safety: Incidence of adverse events | approximately 13 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (1):
- Marlton, New Jersey, United States